CLINICAL TRIAL: NCT07299552
Title: Effects of Vitamin D on Salivary Opiorphin Level, Pain Perception and Tooth Movement in Patients Undergoing Fixed Orthodontic Mechanotherapy
Brief Title: Effects of Vitamin D in Patients Undergoing Fixed Orthodontic Mechanotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Gao Lu, Doctor, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/25030319
Record Dates: First submitted 2025-11-20; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Malocclusions
MeSH Terms: conditions — Malocclusion | interventions — Vitamin D; Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Group (Experimental): Participants receive a 1000 IU vitamin D tablet daily for 4 months during orthodontic treatment.
  Interventions: Dietary Supplement: Vitamin D (Calcitriol)
- Placebo Group (Placebo Comparator): Participants receive a placebo (without vitamin D) daily for 4 months during orthodontic treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D (Calcitriol) — Participants receive a 1000 IU vitamin D tablet daily for 4 months during orthodontic treatment. The supplement is provided in tablet form to participants in the experimental group.
  Arms: Vitamin D Group
Other: Placebo — Oral administration of a placebo (look-alike substance without active vitamin D ingredient), taken daily for 4 months during fixed orthodontic mechanotherapy. The placebo is formulated to match the appearance (e.g., shape, color) and dosage form of the vitamin D supplement provided to the experimental group.
  Arms: Placebo Group

SUMMARY:
The goal of this interventional research is to determine the impact of vitamin D intake on substances in saliva, pain, tooth movement, and the density of the bone around teeth in patients during orthodontic treatment. It will compare the effects of vitamin D supplementation with a placebo to clarify its role in the aforementioned aspects of orthodontic care. The main questions it aims to answer are:

How does vitamin D supplementation affect salivary opiorphin levels in patients undergoing fixed orthodontic mechanotherapy at Specialist Hospital Universiti Sains Malaysia? What is the impact of vitamin D supplementation on pain perception during fixed orthodontic mechanotherapy? How does vitamin D supplementation influence the rate and quality of tooth movement in patients undergoing fixed orthodontic mechanotherapy? What is the relationship between salivary opiorphin levels and pain perception in patients supplemented with vitamin D during fixed orthodontic mechanotherapy? How does vitamin D supplementation affect changes in alveolar bone density during fixed orthodontic mechanotherapy? Researchers will provide vitamin D to the experimental group while the control group receives a placebo to see if vitamin D intake has an impact on substances in saliva, pain, tooth movement, and the density of the bone around teeth during orthodontic treatment.

Participants will:

Take vitamin D or a placebo every day for 4 months Visit the clinic once every 4 weeks for checkups and tests Participate in the study for a duration of up to 4 months

ELIGIBILITY:
Inclusion Criteria:

1. Age Range: 18 to 35 years old. This age group is common and suitable for orthodontic treatment. During this period, skeletal remodeling is active, which is conducive to observing tooth movement and related physiological changes. It is also a stage where the regulatory effects of vitamin D on growth, development, and physiological functions are more pronounced.
2. Orthodontic Requirement: Patients diagnosed with Class I malocclusion with extraction of all first premolars in both upper and lower arches, using MBT orthodontic brackets，and recruited from multiple operators.
3. Health Status: Patients should be in good general health, without endocrine system diseases that affect calcium and phosphorus metabolism and bone metabolism (such as hyperthyroidism or hypothyroidism, parathyroid diseases, etc.). They should also have no severe liver or kidney diseases (since abnormal liver and kidney functions can interfere with the activation and metabolism of vitamin D), and no autoimmune diseases (as autoimmune abnormalities may affect the inflammatory response and tissue repair mechanisms, thus interfering with the experimental results).
4. Medication History: Patients who have not taken any medications affecting calcium and phosphorus metabolism (such as bisphosphonates), bone metabolism (such as recombinant human growth hormone or other drugs that promote or inhibit bone growth), and pain perception (such as long-term use of opioid analgesics, antidepressants that affect neurotransmitters) within the past three months are eligible. This ensures that the experiment is not interfered with by external drug factors.

Exclusion Criteria:

1. Oral Local Problems: Patients with uncontrolled acute or chronic oral inflammations are excluded, such as the acute stage of pericoronitis of wisdom teeth, severe gingivitis, or periodontitis in the progressive and destructive stage. Such inflammations can interfere with the reaction of orthodontic teeth to force and pain assessment. Those with oral mucosal lesions that affect the comfort of wearing orthodontic appliances and the stability of the oral microenvironment are also excluded.
2. Systemic Diseases: Besides the aforementioned endocrine, liver and kidney, and autoimmune diseases, patients with severe cardiovascular diseases (who may have difficulty tolerating the stimulation of orthodontic force application and the regular follow-up process), hematological diseases (which affect blood coagulation and tissue repair and increase the risks of orthodontic treatment), malignant tumors (undergoing radiotherapy or chemotherapy that affects systemic metabolism and immunity) are also excluded. These systemic diseases will introduce too many complex variables and affect the observation of the single factor effect of vitamin D.
3. Special Physiological Periods or Conditions: Pregnant or lactating women are excluded because of the significant fluctuations in hormones and the special nutritional requirements of the fetus or infant, which change the pattern of calcium and phosphorus metabolism. Patients with a recent history of major traumas such as fractures, whose bodies are in a critical period of trauma repair and bone metabolism is in a special stress state, are also not suitable for this experiment as it may interfere with the study of normal orthodontic bone remodeling.
4. Poor Compliance: Patients who cannot be guaranteed regular follow-ups, take medications as prescribed, and cooperate with various examinations are excluded. For example, those with mental or psychological disorders that make it difficult to follow the medical plan, or those who are highly mobile and unable to maintain stable and continuous treatment and observation. Excluding such patients ensures the integrity and reliability of experimental data and the smooth progress of the experimental process.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Salivary Opiorphin Levels During Fixed Orthodontic Mechanotherapy | Baseline assessment, followed by checkups every four weeks over the 4-month period
  Quantify salivary opiorphin concentrations using Human Opiorphin enzyme-linked immunosorbent assay(ELISA) Kit （unit: ng/mL）to evaluate changes associated with vitamin D supplementation.
Pain Perception During Fixed Orthodontic Mechanotherapy | Baseline assessment, followed by checkups every four weeks over the 4-month period
  Assess pain intensity and frequency using a validated pain rating scale (e.g., visual analog scale) to determine the effect of vitamin D supplementation.Visual analog scale(VAS) is a validated, self-reported instrument assessing average pain intensity，Possible scores range from 0 (no pain) to 10 (worst possible pain). A clinically significant difference was considered to be a change by 3 points.
Rate of Tooth Movement During Fixed Orthodontic Mechanotherapy | Baseline assessment, followed by checkups every four weeks over the 4-month period
  Measure tooth movement parameters (i.e., Little's Irregularity Index，unit: millimetres [mm]) via intraoral scan models to evaluate the influence of vitamin D supplementation.
Analyze the relationship between salivary opiorphin levels and pain perception in patients supplemented with vitamin D during fixed orthodontic mechanotherapy. | through study completion, an average of 1 year
  Analyze the correlation between salivary opiorphin levels (unit: ng/mL; measurement tool: enzyme-linked immunosorbent assay [ELISA]) and pain perception (unit: score, 0-10; measurement tool: 100-mm visual analog scale [VAS]) in patients supplemented with vitamin D during fixed orthodontic mechanotherapy.
Evaluate the effects of vitamin D supplementation on changes in alveolar bone density during fixed orthodontic mechanotherapy. | Baseline assessment, followed by a final checkup at the end of the 4-month period
  Cone Beam Computed Tomography (CBCT) will be conducted to assess baseline alveolar bone density on the buccal, lingual, mesial, and distal aspects of tooth roots, as well as in specific jaw regions (e.g., condyle, mandibular angle, maxillary sinus floor).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pakar Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No